CLINICAL TRIAL: NCT05033535
Title: Efficacy and Safety of s086 Tablets in the Treatment of Mild to Moderate Essential Hypertension:a Randomized,Double-blind,Placebo-controlled,Multicenter Phase II Clinical Trial
Brief Title: s086 Tablets in the Treatment of Mild to Moderate Essential Hypertension
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shenzhen People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: S086 Treat hypertension
Record Dates: First submitted 2021-08-25; First posted 2021-09-05 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-08

CONDITIONS: Essential Hypertension
MeSH Terms: conditions — Essential Hypertension | interventions — Olmesartan Medoxomil

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- S086 (Experimental)
  Interventions: Drug: Sacubatril Allisartan medoxomil
- Olmesartan medoxomil (Placebo Comparator): S086 PLCEBO
  Interventions: Drug: Olmesartan Medoxomil

INTERVENTIONS:
Drug: Sacubatril Allisartan medoxomil — Sacubatril Allisartan medoxomil ：A randomized, double-blind, placebo and positive drug parallel controlled, multi-center phase II clinical study on the effectiveness and safety of treating mild and moderate essential hypertension
  Arms: S086
Drug: Olmesartan Medoxomil — Efficacy for lowering blood pressure of Olmesartan medoxomil
  Other Names: Efficacy for lowering blood pressure of Olmesartan medoxomil
  Arms: Olmesartan medoxomil

SUMMARY:
Efficacy and Safety of s086 Tablets in the Treatment of Mild to Moderate Essential Hypertension:a Randomized,Double-blind,Placebo-controlled,Multicenter Phase II Clinical Trial

ELIGIBILITY:
Inclusion Criteria:

* For mild to moderate essential hypertension
* not receiving treatment or being treated with antihypertensive drugs (single drug or combination therapy of two drugs, including compound preparations containing 2 drug components)
* not receiving treatment (newly diagnosed Essential hypertension or a history of hypertension but not taking any antihypertensive drugs at least 4 weeks before screening), during the screening period (V1) and before randomization (V4), the mean sitting systolic blood pressure (msSBP) ≥ 150mmHg and <180mmHg;
* patients who are receiving antihypertensive drugs (treated with antihypertensive drugs within 4 weeks before screening), at the end of the wash period (V2), must meet the average sitting systolic blood pressure ≥140mmHg and <180mmHg; before randomization (V4), the average sitting systolic blood pressure must be ≥150mmHg and <180mmHg;
* the patient's average sitting systolic blood pressure before randomization (V4) must be the difference between the previous average sitting systolic pressure (at the end of the washing period (V2)) ≤15mmHg; voluntarily participate in the trial and sign an informed consent form.

Exclusion Criteria:

* Have a history of allergies to relevant components of the test drug, known or suspected to be allergic to S086, sacubatril, valsartan sodium or olmesartan medoxomil and related drugs (ARB, ACEI, and renin inhibitors);
* currently in pregnancy, breastfeeding Female subjects whose pregnancy or pregnancy tests are positive; or those whose subjects or their partners cannot guarantee effective contraception during the trial period (acceptable methods of contraception: true abstinence; intrauterine contraceptive devices; barrier contraceptives; or partners accepted Sterilization surgery. Unacceptable contraceptive methods: periodic abstinence, such as contraception based on calendar, ovulation, symptomatic body temperature);
* or those who have a childbirth plan within 6 months after the end of the trial;
* have a history of drug abuse or alcohol abuse within 6 months before screening History: Participated in any drug or medical device or other clinical trial within 3 months before screening, or participated in any drug or medical device or other clinical trial during the planned trial or within 3 months after the end of the trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
sitting systolic blood pressure (msSBP) | 8 weeks after baseline
  sitting systolic blood pressure (msSBP) at the 8th weekend from baseline

SECONDARY OUTCOMES:
sitting Diastolic blood pressure (msDBP) | 8 weeks after baseline
  sitting Diastolic blood pressure (msDBP) at the 8th weekend from baseline
Compliance rate | 8 weeks after baseline
  Compliance rate of pressure reduction at the 8th weekend

CONTACTS AND LOCATIONS:
Locations (1):
- Shenzhen People' S Hospital, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No